CLINICAL TRIAL: NCT04511533
Title: SINGLE ARM STUDY TO EVALUATE THE SAFETY OF DACOMITINIB FOR THE FIRST-LINE TREATMENT OF PARTICIPANTS IN INDIA WITH METASTATIC NON-SMALL CELL LUNG CANCER WITH EPIDERMAL GROWTH FACTOR RECEPTOR (EGFR)-ACTIVATING MUTATIONS
Brief Title: Dacomitinib for Treatment of Patients in India With Metastatic Non Small Cell Lung Cancer With EGFR Activating Mutations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A7471064
Record Dates: First submitted 2020-07-30; First posted 2020-08-13 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Non Small Cell Lung Cancer
Keywords: Dacomitinib; Metastatic Non Small Cell Lung Cancer; EGFR-activating mutations; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): The recommended dosage of dacomitinib is 45 mg taken orally once a day at approximately the same time each day, until disease progression, participant refusal/lost to follow-up, or unacceptable toxicity occurs.
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib — Dacomitinib is a kinase inhibitor indicated for the first line treatment of patients with metastatic NSCLC with EGFR exon 19 deletion or exon 21 L858R substitution mutations.
  Other Names: DACOPLICE

SUMMARY:
This is a Phase 4, open label, single arm, multi-center, prospective clinical trial of dacomitinib that will be performed in India. This study will enroll a sufficient number of participants to ensure that 100 participants are treated with dacomitinib. The primary objective of this study is to assess the safety and tolerability of dacomitinib. The secondary objective is to evaluate antitumor activity of dacomitinib by objective response rate and duration of response.

DETAILED DESCRIPTION:
This is a Phase 4, open label, single arm, multi-center, prospective clinical trial of dacomitinib that will be performed in India. This study will enroll a sufficient number of participants to ensure that 100 participants are treated with dacomitinib. The primary objective of this study is to assess the safety and tolerability of dacomitinib. The secondary objective is to evaluate antitumor activity of dacomitinib by objective response rate and duration of response. Drug administration: Dacomitinib will be supplied by Pfizer and administered in accordance with the India Local Product Document (LPD). The recommended dosage of dacomitinib is 45 mg taken orally once a day at approximately the same time each day, until disease progression, participant refusal/lost to follow-up, or unacceptable toxicity occurs.

STUDY PROCEDURES:

Screening: Participants will be screened within 28 days prior to first dosing of dacomitinib to confirm that they meet the eligibility criteria for the study.

Follow-up Visit: All participants will return to the study site up to 28 days after the last dose of study drug administration for assessment of potential AEs, recording of concomitant treatment use and to confirm appropriate contraception usage.

ASSESSMENTS Tumor Assessments: Tumor assessments will include all known or suspected disease sites. Computerized tomography (CT) or Magnetic resonance imaging (MRI) scans of Chest Abdomen and Pelvis and MRI of the brain will be performed at Screening and repeated every 12 weeks ±1 week until the end of treatment. For all tumor assessments, the method of assessment that was used at Screening will be used throughout the study. Tumor assessment will be repeated at the end of treatment if more than 6 weeks have passed since the last evaluation. Assessment of response will be made using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Confirmation of response will be required ≥4 weeks after initial response is observed.

Safety Assessments: The following parameters will be assessed - Physical examination, vital signs, Eastern Cooperative Oncology Group Performance score (ECOG PS), safety lab data, 12 lead electrocardiogram (ECG). Unscheduled clinical laboratory measurements may be obtained at any time during the study to assess any perceived safety concerns.

Adverse event reporting: All observed or volunteered AEs regardless of treatment group or suspected causal relationship to the investigational product(s) will be reported as per regulatory requirements.

End of Study: The end of study is defined as 1 year after the last participant first visit (LPFV) date in the study. At the end of study, participants who are on treatment and benefiting from dacomitinib treatment will be switched to commercially available dacomitinib if considered appropriate by the investigator, as soon as feasible.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of histologically or cytologically confirmed diagnosis of metastatic NSCLC with EGFR activating mutations as detected by an appropriate test.
2. No prior treatment with systemic therapy and EGFR/Other Tyrosine Kinase Inhibitors (TKIs) for metastatic NSCLC.
3. Participants with asymptomatic Central Nervous System (CNS) metastases (including participants controlled with stable or decreasing steroid use within the last 2 weeks prior to study entry) will be eligible.
4. Age >=18 years.
5. ECOG PS of 0-2.
6. Adequate . hematologic, renal, liver function: ANC >= 1000/mm3; Platelets>=50000/mm3; Hb >=8 g/dL; est. Cr.Cl >=30 mL/min; Total serum bilirubin <1.5 × ULN; AST,ALT <=2.5 × ULN; (<=5.0 × ULN, if liver metastases).
7. Acute effects of any prior therapy resolved to baseline severity or to Common Terminology Criteria for Adverse Events (CTCAE) Grade <1 except for AEs that in the investigator's judgment do not constitute a safety risk for the participant.
8. Serum or urine pregnancy test (for females of childbearing potential) negative at Screening.

Exclusion Criteria:

1. Any evidence of mixed histology that includes elements of small cell or carcinoid lung cancer.
2. Any other mutation other than exon 19 deletion or L858R in exon 21, with or without the presence of the exon 20 T790M mutation.
3. Radiation therapy (except palliative to relieve bone pain) within 2 weeks of study entry. Prior irradiation to >25% of the bone marrow.
4. Major surgery within 4 weeks prior to first dose of dacomitinib. Minor surgical procedures (eg, port insertion) are not excluded, but sufficient time should have passed for adequate wound healing.
5. Known prior or suspected severe hypersensitivity to dacomitinib or any component of its formulation.
6. History or known presence of interstitial fibrosis, interstitial lung disease, pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, obliterative bronchiolitis, and pulmonary fibrosis.
7. Other severe acute or chronic medical or psychiatric condition, that may interfere with the interpretation of study results and, would make the participant inappropriate for entry into this study.
8. Evidence of active malignancy (other than current NSCLC) within the last 3 years prior to first dose of dacomitinib.
9. Breastfeeding female participants.
10. Pregnant female participants; male participants able to father children and female participants of childbearing potential who are unwilling or unable to use contraception method per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- India (15):
  - The Gujarat Cancer and Research Institute, Ahmedabad, Gujarat
  - Hemato Oncology Clinic Ahmedabad Pvt. Ltd, Ahmedabad, Gujarat
  - Gujarat Hospital - Gastro & Vascular Centre, Surat, Gujarat
  - Unity Trauma Center And ICU (Unity Hospital ), Surat, Gujarat
  - Artemis hospital, Gurugram, Haryana
  - National Cancer Institute, Nagpur, Maharashtra
  - Apex Wellness Hospital, Nashik, Maharashtra
  - Grant Medical Foundation, Ruby Hall Clinic, Pune, Maharashtra
  - Sahyadri Clinical Research and Development Center, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Bhaktivedanta Hospital and Research Institute, Thane, Maharashtra
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, National Capital Territory of Delhi
  - Yashoda Hospital, Hyderabad, Telangana State
  - Netaji Subhas Chandra Bose Cancer Hospital, Kolkata, West Bengal
  - Tata Medical Center, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A7471064

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 106 participants were screened, 5 participants were screen failures, 101 participants were enrolled and assigned to treatment and all of them were treated.
Groups:
- Dacomitinib: Participants with metastatic non-small cell lung carcinoma (NSCLC) with epidermal growth factor receptor (EGFR) mutations received a starting dose of dacomitinib 45 mg once daily in each cycle of 28 days, until disease progression, participant refusal/lost to follow-up, or unacceptable toxicity occurred. The maximum treatment duration was approximately 107.3 weeks.
Period: Treatment
Arm/Group | Dacomitinib
Started | 101
Completed | 21
Not Completed | 80
Not completed — Other | 2
Not completed — Withdrawal by Subject | 11
Not completed — Death | 5
Not completed — Physician Decision | 1
Not completed — Progressive Disease | 61
Period: Follow-Up
Arm/Group | Dacomitinib
Started | 96 (5 Participants died during the treatment phase, therefore did not enter the follow-up phase.)
Completed | 78
Not Completed | 18
Not completed — Other | 7
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 2
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants enrolled and treated in the study.
Arm/Group | Dacomitinib
Number analyzed (Participants) | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 75
  >=65 years | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.95 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 101
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-Causality and Treatment-Related Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Relatedness to study drug was assessed by the investigator. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to approximately 107.3 weeks that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the first dose of study treatment up to 28 days after the last dose of study treatment (maximum treatment duration: 107.3 weeks)
Population: All participants who received at least 1 dose of dacomitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib
Number analyzed (Participants) | 101
Participants
  Number of Participants with all-causality TEAEs | 94
  Number of Participants with all-causality SAEs | 16
  Number of Participants with treatment-related TEAEs | 92
  Number of Participants with treatment-related SAEs | 7

2. Secondary Outcome: Overall Response Rate (ORR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 Based on Investigator Assessment
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST. Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. Per RECIST v1.1: CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. Stable disease was defined as not qualifying for CR, PR, Progressive Disease.
Time Frame: From time of first dose until disease progression, death or initiation of a new anticancer therapy, whichever occurs first, assessed for up to 26 months
Population: All participants who received at least 1 dose of dacomitinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dacomitinib
Number analyzed (Participants) | 101
Percentage of participants | 50.5 [40.9 to 60.0]

3. Secondary Outcome: Duration of Response (DOR) as Per RECIST Version 1.1 Based on Investigator Assessment
Description: DOR: time from first documented occurrence of response (PR or CR) until date of first documented PD or death due to underlying cancer. RECIST 1.1. CR: disappearance of all non-nodal target lesions and of all non-target lesions. In addition, any pathological lymph nodes assigned as target lesions/ non-target lesions must have a reduction in short axis to <10 mm. PR: at least a 30% decrease in sum of diameter of all target lesions, taking as reference baseline sum of diameters. PD: at least a 20% increase in sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm^2. Unequivocal progression of existing non-target lesions. Appearance of new lesions. Participants with no PD and were still alive, were censored at last adequate tumor assessment. Kaplan-Meier method was used for DOR analysis.
Time Frame: From time of first tumor response until disease progression, death or initiation of a new anticancer therapy, whichever occurs first, assessed for up to 26 months
Population: All participants who received at least 1 dose of dacomitinib. DOR was only for the subset participants with an objective response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dacomitinib
Number analyzed (Participants) | 51
Months | 11.1 [8.3 to 16.6]

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment up to a minimum of 28 days after the last dose of study treatment (maximum treatment duration: 107.3 weeks)
Arm/Group | Dacomitinib
All-Cause Mortality (participants affected / at risk) | 9/101
Serious Adverse Events (participants affected / at risk) | 16/101
Other Adverse Events (participants affected / at risk) | 93/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dacomitinib (N=101)
Asthenia (General disorders) | 1
Death (General disorders) | 2
Disease progression (General disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
COVID-19 (Infections and infestations) | 2
COVID-19 pneumonia (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Cardiac arrest (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Blood creatinine increased (Investigations) | 1
SARS-CoV-2 test positive (Investigations) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dacomitinib (N=101)
Anaemia (Blood and lymphatic system disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 52
Mouth ulceration (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 7
Chest pain (General disorders) | 7
Mucosal inflammation (General disorders) | 11
Pyrexia (General disorders) | 8
Paronychia (Infections and infestations) | 26
Weight decreased (Investigations) | 35
Decreased appetite (Metabolism and nutrition disorders) | 10
Hypokalaemia (Metabolism and nutrition disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 25
Pruritus (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT04511533/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT04511533/SAP_001.pdf